CLINICAL TRIAL: NCT04054791
Title: Endonasal Dacryocystorhinostomy: Prospective Study of the Evolution of the Stoma Size
Brief Title: Endonasal Dacryocystorhinostomy and Evolution of the Stoma Size
Acronym: EndoDCRevol
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-10Obs-CHRMT
Record Dates: First submitted 2019-08-08; First posted 2019-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Endonasal Dacryocystorhinostomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Dacryocystorhinostomy (DCR) is a procedure of choice for nasolacrimal duct obstruction. Endonasal procedures for DCR were described as early as 1893 by Caldwell. However, external DCR was practiced more commonly because of better visualization of anatomic features. The miniaturization of surgical instruments and close partnership between ophthalmologist and otorhinolaryngologist had led to a renewal of endonasal approach.

The main objective of the study is to show the evolution of stoma size after endonasal DCR and validate the direct measurement of mucous orifice. It will also allow determining if the stoma evolution size may be a predictive factor for operational effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Patient with chronic epiphora or chronic dacryocystitis

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had chronic epiphora or chronic dacryocystitis.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Evolution of the stoma size | Month 12
  Measurement of the stoma size by endonasal photography

SECONDARY OUTCOMES:
Mucous orifices size | Month 2
  Measurement of the osteotomy orifices size from photography
Ratio of patients for whom the operation is a success | Month 12
  A success corresponds to the complete disappearance of epiphora symptomatology, on the contrary, a failure equals to the persistence of tearing or a recurrence of dacryocystitis